CLINICAL TRIAL: NCT01576185
Title: Development of Pediatric Acute Myeloid Leukemia Xenograft Models for the Testing of Targeted Therapeutic Agents
Brief Title: Developing and Treating a Mouse Model of Acute Myeloid Leukemia Using Tissue Samples From Younger Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML12B8; NCI-2012-00724 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-AAML12B8 (Other: Children's Oncology Group); CDR0000730390 (Other: Clinical Trials.gov)
Record Dates: First submitted 2012-04-11; First posted 2012-04-12 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Childhood Acute Myeloid Leukemia/Other Myeloid Malignancies
MeSH Terms: interventions — quizartinib; Sorafenib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational (xenograft models): Human acute myeloid leukemia cells are injected into NSG mice. Mice are then treated with sorafenib or quizartinib via gavage once daily for 28 days. Peripheral blood and tissue samples are collected biweekly or weekly and analyzed for the presence of human CD45+ and CD33+ cells by quantitative flow cytometry.
  Interventions: Other: laboratory biomarker analysis; Drug: quizartinib; Drug: sorafenib tosylate

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies
Drug: quizartinib — Via gavage
  Other Names: AC220; class III receptor tyrosine kinase inhibitor AC220
Drug: sorafenib tosylate — Via gavage
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN

SUMMARY:
These laboratory trial studies the development and treatment of a mouse model for acute myeloid leukemia (AML) using samples from younger patients with AML. Studying tissue samples from patients with cancer in the laboratory may help doctors learn more about cancer and how well patients will respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the rate of engraftment of pediatric FMS-Like Tyrosine Kinase-3 (FLT3)-internal tandem duplication (ITD) acute myeloid leukemia (AML) samples in NOD scid gamma (NSG) mice.

II. To determine the efficacy of treatment of FLT3-ITD xenografts with tyrosine kinase inhibitors.

OUTLINE:

Human acute myeloid leukemia cells are injected into NSG mice. Mice are then treated with sorafenib or quizartinib via gavage once daily for 28 days. Peripheral blood and tissue samples are collected biweekly or weekly and analyzed for the presence of human CD45+ and CD33+ cells by quantitative flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* Cryopreserved human AML samples

  * FLT3-ITD samples with high allelic ratios

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cryopreserved human AML samples FLT3-ITD samples with high allelic ratios
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Engraftment ratio of human AML cells to murine cells | Up to 9 months
  We will measure total leukemic burden from harvested femurs, tibias, and spleen by quantitative flow cytometry, estimate engraftment, and describe 95% confidence intervals. The total AML cell count of the control and treatment cohorts will be compared using an analysis of variance (ANOVA) test.
Efficacy of sorafenib or quizartinib to inhibit AML proliferation in vivo | Up to 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Tasian, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States